CLINICAL TRIAL: NCT06933927
Title: Evaluation of Gingival Health and Bacterial Adhesion of Bioflx Crowns Compared to Zirconia Crowns on Primary Molars: A Randomized Clinical Trial
Brief Title: Comparative Evaluation of Gingival Health and Bacterial Adhesion in Bioflx vs. Zirconia Crowns on Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Ahmed Abdelrazig Mohammed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EGHBA-BFXZRC-PM-2025
Record Dates: First submitted 2025-04-10; First posted 2025-04-18 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Carious Primary Molars

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bioflex crowns (Experimental): Bioflx Crowns (BFCs) the first flexible, durable, and esthetic preformedcrown for primary molars .BFCs are monochromatic, metal-free, tooth-colored crowns used in the medical device industry having high strength, flexibility, and durability. These crowns are autoclavable and are similar to SSC in tooth preparation. Additionally, they offer a cost benefit compared to zircon crowns
  Interventions: Other: (Group A: Bioflx crowns)
- Zirconia crowns (Experimental): zirconia crowns are frequently chosen as a comparator due to their established clinical performance and favorable biological properties. Studies have demonstrated that zirconia crowns exhibit lower bacterial adhesion, particularly of Streptococcus mutans, compared to stainless steel crowns (SSCs). highly polished and smooth surface of zirconia, which minimizes plaque accumulation and subsequent gingival inflammation.
  Interventions: Other: (Group B) : Preformed Zirconia crown

INTERVENTIONS:
Other: (Group A: Bioflx crowns) — Minimal preparation will be required due to their flexural adaptability:1. Choose an appropriately sized Bioflex (Nusmile) crown of similar size to the mesiodistal width.2. The tooth will be prepared using a flame stone for occlusal reduction by 1-1.5 mm, including the central groove .3Proximal preparation will be around 0.5 mm, by using a fine, long, tapered diamond stone to cut interproximal slices mesially and distally.4. The crown will be placed with a snug fit and cemented using glass ionomer
  Arms: Bioflex crowns
Other: (Group B) : Preformed Zirconia crown — 1. Size Determination can be achieved by holding a crown up to the existing tooth or, if available, using digital x-ray measurements to match the patient's interproximal width to the corresponding crown size.2. OcclusalPerform an occlusal reduction of about 1.5-2 mm, ensuring adequate space for the crown material. 3. Axial ReductionReduce the buccal and lingual surfaces uniformly, ensuring the removal of any prominent buccal bulges to allow for a passive crown fit. 4. Interproximal ReductionClearance: Ensure sufficient interproximal space by removing enough tooth structure to allow the crown to seat without interference.5. Subgingival PreparationMargin Placement: Extend the preparation subgingivally by approximately 2 mm to achieve optimal crown retention and aesthetics. This involves removing the chamfer margin at the tissue level and ensuring a smooth transition from the root to the coronal tooth structure
  Arms: Zirconia crowns

SUMMARY:
The goal of this clinical trial is to evaluate the Evaluation of Gingival Health and Bacterial Adhesion of Bioflx Crowns Compared to Zirconia Crowns on Primary Molars of Bioflx crowns compared to zirconia crowns in the restoration of primary molars. The main question[s] it aims to answer is there are the differences in bacterial adhesion and gingival health between bioflx and zirconia crowns The study will also assess the clinical performance of both types of crowns in terms of bacterial adhesion , child and parents satisfaction,as well as preparation time.

DETAILED DESCRIPTION:
Dental caries is an oral disease most ubiquitous among children, characterized by a series of demineralization and remineralization cycles. If left untreated, it can progress to cavitated lesions. Usually, the familiar method of managing multi-surface carious lesions in primary teeth with stainless steel crowns .Streptococcus mutans is considered to be the main colonizer and primary etiological factor in caries progression as it stimulates the production of glucans from the food substrates. Research has indicated that S. mutans can be isolated from plaque samples. Consequently the long-term success of a restored tooth is significantly affected by the adhesion of S. mutans to the preformed crowns.Bacterial adhesion on zirconia are sparse. An in vitro study reported the initial bacterial adhesion on the surface of zirconia to be less compared with resins. When a primary tooth is restored with a full-coverage restoration, it establishes a fresh environment conducive to microbial adhesion. Bioflx Crowns the first flexible, durable, and esthetic preformedcrown for primary molars .BFCs are monochromatic, metal-free, tooth-colored crowns used in the medical device industry having high strength, flexibility, and durability. These crowns are autoclavable and are similar to SSC in tooth preparation. Additionally, they offer a cost benefit compared to zircon crowns,

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 4-8 years.
2. decayed in primary molars require full-coverage crowns.
3. No history of systemic diseases affecting oral health.
4. Cooperative children.

Exclusion Criteria:

-patients with severe medical conditions, badly decayed in primary molars and trauma.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Gingival Health | 6 months
  plaque index using Silness& Löe plaque index:0 - 3 0: no plaque.1: film at gingival margin.2: moderate accumulation.3: abundance of plaque.
Gingival health | 6 months
  Gingival index using Löe& Silness :0 - 3 0: healthy gum.1: mild discoloration and edematous gingiva, no bleeding on probing.2: red oedematous and shiny gingiva,bleeding on probing.3: red oedematous and ulceration gingiva, spontaneous bleeding.

SECONDARY OUTCOMES:
Bacterial adhesion | 2 weeks
  Method of measurement : by( Mitis salivarius agar) Unit of measurement :Colony-formingunits.
child and parental satisfaction | 6 months
  5-Point likert's scale / Questionnaire.
  1. Very Happy.2. Happy.3. Neither.4. Unhappy.5. Very Unhappy.
Preparation time | 6 months
  Method of measurement : stop watch Unit of measurement : minutes

CONTACTS AND LOCATIONS:
Overall Officials: Manal Ahmed Elsheikh, PHD, Study Director — Cairo University; Shaimaa Mohamed Sabry mostafa, PHD, Study Director — Cairo University
Locations (1):
- Faculty of dentistry cairo university, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Background] Patil AS, Jain M, Choubey S, Patil M, Chunawala Y. Comparative evaluation of clinical success of Stainless Steel and Bioflx crowns in primary molar - A 12 month split mouth prospective randomized clinical trial. J Indian Soc Pedod Prev Dent. 2024 Jan 1;42(1):37-45. doi: 10.4103/JISPPD.JISPPD_484_23. Epub 2024 Apr 15. PMID 38616425
- [Background] Bin AlShaibah WM, El-Shehaby FA, El-Dokky NA, Reda AR. Comparative study on the microbial adhesion to preveneered and stainless steel crowns. J Indian Soc Pedod Prev Dent. 2012 Jul-Sep;30(3):206-11. doi: 10.4103/0970-4388.105012. PMID 23263423